CLINICAL TRIAL: NCT00310830
Title: Randomized, Placebo-controlled, Double-blind, Multicenter, Parallel Group Study to Assess the Efficacy, Safety and Tolerability of Bosentan in Patients With Symptomatic Pulmonary Arterial Hypertension Associated With Sickle Cell Disease
Brief Title: Efficacy and Safety of Bosentan in Sickle Cell Disease (SCD) Patients With Pulmonary Arterial Hypertension (PAH)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Slow enrollment
Sponsor: Actelion (Industry)
Responsible Party: Sebastien Roux, MD, Actelion
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AC-052-368; ASSET-1; NCT00307359 (obsolete NCT alias)
Record Dates: First submitted 2006-04-03; First posted 2006-04-05 (Estimated); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Pulmonary Hypertension
Keywords: Pulmonary Arterial Hypertension; Pulmonary hypertension; Sickle Cell Disease; Sickle cell anemia; ASSET; ASSET-1
MeSH Terms: conditions — Hypertension, Pulmonary; Pulmonary Arterial Hypertension; Anemia, Sickle Cell | interventions — Bosentan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- 1 (No Intervention)
- 2 (Experimental)
  Interventions: Drug: Bosentan

INTERVENTIONS:
Drug: Bosentan — Oral, Initial dose: 62.5 mg b.i.d. for 4 weeks, maintenance dose: 125 mg b.i.d.
  Arms: 2

SUMMARY:
The study will assess the effect of bosentan on pulmonary vascular resistance and exercise capacity in sickle cell disease (SCD) patients diagnosed with pulmonary arterial hypertension. It consists of 3 phases: Screening, Treatment and Follow-up. During the Screening visit, the study doctor will decide if patients meet the study requirements. All potential patients will have a diagnosis of increased pulmonary artery pressures that is shown by right heart catheterization conducted shortly prior to start of study treatment. Patients will be asked to perform exercise capacity test (walking as far as possible for 6 minutes). Following the Baseline visit, the treatment phase consists of 4 additional clinic visits during which the good and bad effects of the drug are reviewed and exercise capacity test will be repeated. Patients will be treated for 16 weeks. Blood samples will be collected every month, or more often, if needed. At the end of the study, patients will be asked to repeat the right heart catheterization and exercise capacity test. After completion of the study, patients will have the option of enrolling in a long-term follow-up study where all patients will receive active drug. Patients electing not to participate in the extension study will be followed up for safety assessments for about 28 days after the end of the study treatment.

ELIGIBILITY:
Inclusion Criteria: Screening Criteria:

1. Males or females ≥ 12 years of age with a documented history of SCD
2. Patients with symptomatic PAH associated with shortness of breath
3. Patients with tricuspid regurgitation jet (TRJ) velocity of > 2.9 m/sec based on echo/Doppler conducted within 6 months prior to randomization and not during SCD crisis
4. Signed written informed consent is obtained from the patient or patient's parent/legal representative prior to initiation of any study related procedure

Inclusion Criteria:

1. Patients with hemoglobin (Hb) SS or Hb S/β0 genotype and with Hb A ≤ 10%
2. Six-minute walk test (6MWT) distance ≥ 150 m and ≤ 450 m
3. PAH confirmed by right heart catheterization (RHC) performed at the study site within 3 months of the randomization visit and defined as:

   * Mean pulmonary arterial pressure (mPAP) ≥ 25 mmHg
   * Pulmonary capillary wedge pressure (PCWP) ≤ 15 mmHg measured by RHC or left ventricular end diastolic pressure (LVEDP) ≤ 15 mmHg measured by left heart catheterization, if PCWP measurement is not reliable
   * Pulmonary vascular resistance (PVR) at rest ≥ 160 dyn.sec/cm5
4. Women of childbearing potential must have a negative result on their serum pregnancy test and use reliable methods of contraception during study treatment and for 3 months after study treatment termination

Exclusion Criteria:

1. Left ventricular ejection fraction < 40% (echo/Doppler)
2. Systolic blood pressure < 85 mmHg
3. Uncontrolled hypertension with systolic blood pressure >160 mmHg and/or diastolic blood pressure > 100 mmHg
4. Forced expiratory volume in 1 second divided by forced vital capacity (FEV1/FVC) < 0.5
5. Total lung capacity (TLC) < 50% of normal predicted value
6. Significant cardiac disease: ischemic, valvular, constrictive
7. Hemoglobin concentration < 6.0 g/dL at the time of randomization
8. Acute liver disease
9. Evidence of cirrhosis or portal hypertension on a liver ultrasound or biopsy
10. ALT ≥ 2 times upper limit of normal (ULN) and/or albumin < 2.8 g/dL
11. Acute or chronic impairment (other than dyspnea), limiting the ability to comply with study requirements (in particular with 6MWT), e.g., angina pectoris, intermittent claudication, symptomatic hip osteonecrosis
12. Vaso-occlusive crisis (VOC) or acute chest syndrome (ACS) within 2 weeks of randomization or more than 12 VOC and/or ACS within the last 12 months
13. Blood transfusion within 4 weeks prior to randomization
14. Illness with a life expectancy shorter than 6 months
15. HIV with opportunistic infection
16. Psychotic, addictive, or other disorder limiting the ability to provide informed consent or to comply with study requirements
17. Pregnant or lactating women
18. Recently started (< 8 weeks prior to randomization) or planned, exercise-based cardio-pulmonary rehabilitation program
19. Bone marrow transplantation
20. Treatment or planned treatment with another investigational drug within 3 months prior to randomization
21. Treatment for pulmonary hypertension with an endothelin receptor antagonist, a phosphodiesterase-5 inhibitor, prostanoids (excluding acute administration during a catheterization procedure to test vascular reactivity) within 3 months prior to randomization or with L-arginine within 1 week prior to randomization
22. Treatment with calcineurin-inhibitors (e.g., cyclosporine A and tacrolimus), sirolimus, fluconazole, amiodarone, miconazole and glibenclamide (glyburide) within 1 week prior to randomization
23. Known hypersensitivity to bosentan or any of its excipients

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2006-03; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Change from Baseline to End of Study in 6MWT distance. A mean difference from placebo of at least 35 m is considered clinically relevant. | 16 weeks

SECONDARY OUTCOMES:
Time to clinical worsening from Baseline to EOS. | 16 weeks

REFERENCES:
- [Derived] Barst RJ, Mubarak KK, Machado RF, Ataga KI, Benza RL, Castro O, Naeije R, Sood N, Swerdlow PS, Hildesheim M, Gladwin MT; ASSET study group*. Exercise capacity and haemodynamics in patients with sickle cell disease with pulmonary hypertension treated with bosentan: results of the ASSET studies. Br J Haematol. 2010 May;149(3):426-35. doi: 10.1111/j.1365-2141.2010.08097.x. Epub 2010 Feb 17. PMID 20175775
- See also: A web site with information for patients about the disease and treatment options — http://www.sicklecelldisease.org/
- See also: A newsletter and information web site — http://www.SCInfo.org